CLINICAL TRIAL: NCT02754869
Title: Post-Hoc Analysis of Dynamic Magnetic Resonance Sequences to Establish Descriptive Metrics for Small Bowel Motility in Vivo
Brief Title: Magnetic Resonance Imaging Assessment of Small Bowel Motility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 11/0307
Record Dates: First submitted 2016-02-23; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2015-11

CONDITIONS: Motility Disorder of Intestine

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Control Subject-Drug Study: The first part of this investigation is an interventional blinded cross over study with two dosing dates spread at least one week apart. Each volunteer will receive baseline scans before drug/placebo which will be used to assess intra---patient variation over the two study dates after which the drug or saline placebo will be administered with each volunteer acting as their own control to assess software ability to quantify changes in bowel motility.
- Dysmotility Subjects-Drug Study: The second component of this study will be exactly the same for the participants with dysmotility except the time to repeat scan will be reduced with a follow up time aimed at around 1---3 days reducing patient time off medication
- Reference Range Study: The third component of this study will assess basal small bowel motility in larger numbers of healthy controls, dysmotility subjects and irritable bowel syndrome to establish reference ranges to inform future clinical investigations and guide clinical decision making using global motility scoring. Each scan will last around 20 minutes and will not involve follow up or use of pharmaceutical agents.
- Desmotility Reversibility Study: The fourth component of the study will assess small bowel motility in a cohort of Crohns disease patients will small bowel disease before and 11---16 weeks after starting anti TNF alpha therapy, or undergoing endoscopic dilatation of a small bowel stricture. Each scan will last around 45 minutes

SUMMARY:
This project involves the development, validation and application of a novel test using MRI to assess gastrointestinal motility a vital process that mixes the contents of our digestive tract. This process frequently becomes deranged in conditions like chronic constipation, Parkinson's and Crohn's disease.

DETAILED DESCRIPTION:
Gastrointestinal motility refers to the contractile actions in the gut that serve to mix our food and propel it through out digestive tract. Although known to be involved in a range of conditions like chronic constipation, Parkinson's and Crohn's disease, investigator have never had effective tests with which to study the process. Advances in medical imaging technologies now make it possible to both see and quantify this process non-invasively using MRI. In this study the investigator first of all validate that our MRI based analysis is robust and valid, producing predictable results against range of known stimuli. The investigator then apply the technique to a cohort of participants with Chronic Intestinal Pseudo-Obstruction. These participants are known to have hypo-motile small bowels and demonstration with our MRI technique would serve as further validation. The investigator also investigate two cohorts of people with and without gastrointestinal diseases to better understand how the technique may work in the clinical setting.

By the end of this project The investigator will have generated robust initial evidence to validate our MRI technique and clinical data to inform use further research.

ELIGIBILITY:
Inclusion Criteria:

ELIGIBILITY CRITERIA - CONTROL SUBJECTS DRUG STUDY:

* Adult (>16 years)
* Body Mass Index within the range of (18---25)

ELIGIBILITY CRITERIA - DYSMOTILITY SUBJECTS DRUG STUDY:

* Adult patients (>16 years) 2
* Dysmotility diagnosis including CIPO
* Body Mass Index within the range of (18---35)

ELIGIBILITY CRITERIA - REFERENCE RANGE STUDY (NORMAL PARTICIPANTS):

• Adult (>16 years)

ELIGIBILITY CRITERIA - REFERENCE RANGE STUDY (DYSMOTILITY/IBS):

* Adult patients (>16 years)
* Dysmotility, CIPO or IBS diagnosis

ELIGIBILITY CRITERIA - DYSMOTILITY REVERSIBILITY STUDY:

* Adult (>16 years)
* Known small bowel Crohn's disease starting anti TNF alpha medication or undergoing endoscopic small bowel stricture dilatation.

Exclusion Criteria:

EXCLUSION CRITERIA - CONTROL SUBJECTS DRUG STUDY:

* Any contraindications to MRI scans (e.g. Implanted cardiac pacemaker, defibrillator device)
* Inability to give consent
* Treatment for any chronic illness
* Use of laxatives, anti---diarrhoeals or any drugs affecting GI motility (including NSAIDs) prohibited within one week of the scan.
* Cardiac symptoms (palpitations).
* Abnormal GI symptoms (eg. constipation, diarrhea, bloating, pain) as per the Rome III criteria for Irritable Bowel Syndrome
* Pregnancy
* Asthma EXCLUSION CRITERIA - DYSMOTILITY SUBJECTS DRUG STUDY: (18) Version 4.1
* Any contraindications to MRI scans (e.g. Implanted cardiac pacemaker, defibrillator device)
* Inability to give consent
* Use of laxatives, anti---diarrhoeals or any drugs affecting GI motility (including NSAIDs) prohibited within 1---3 days (or according to half life of drug) of the scan.
* Cardiac symptoms (palpitations).
* Pregnancy
* Asthma

EXCLUSION CRITERIA - REFERENCE RANGE STUDY (NORMAL PARTICIPANTS):

* Any contraindications to MRI scans (e.g. Implanted cardiac pacemaker, defibrillator device)
* Inability to give consent 3. Treatment for any chronic illness
* Use of laxatives, anti---diarrhoeals or any drugs affecting GI motility (including NSAIDs) prohibited within 1---3 days (or according to half life of drug) of the scan.

EXCLUSION CRITERIA - REFERENCE RANGE STUDY (DYSMOTILITY/IBS):

* Any contraindications to MRI scans (e.g. Implanted cardiac pacemaker, defibrillator device)
* Inability to give consent
* Use of laxatives, anti---diarrhoeals or any drugs affecting GI motility (including NSAIDs) prohibited within 1---3 days (or according to half life of drug) of the scan.

EXCLUSION CRITERIA - DYSMOTILITY REVERSIBILITY STUDY:

* Any contraindications to MRI scans (e.g. Implanted cardiac pacemaker, defibrillator device)
* Inability to give consent
* Use of laxatives, anti---diarrhoeals or any drugs affecting GI motility (including NSAIDs) prohibited within 1---3 days (or according to half life of drug) of the scan.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers on the placebo---controlled drug study using neostigmine will be recruited from UCL staff and student population by internal advertisement. Patients with CIPO and (13) Version 4.1 dysmotility will be identified from patient records held in the gastroenterology departments at UCL and Queen Mary's University London.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2011-02; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
To establish the reproducibility of software quantified small bowel motility in normal individuals using processed MRI derived dynamic small bowel sequences. | 7 years
To assess the ability of the software to detect changes in small bowel motility after provocation with a known pro or anti-kinetic agent in normal individuals | 7 years
To evaluate the variation in software quantified small bowel motility according to the positioning of the image slice in the abdomen during data acquisition. | 7 years
To compare dysmotility patients motility to that of normal controls with and in the absence of pro---kinetic agent. | 7 years
To establish basal bowel motility reference ranges in a larger cohort of control, dysmotility and irritable bowel syndrome subjects. | 7 years
To assess the reversibility of dysmotility after treatment of the primary underlying condition, if known | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Taylor, Principal Investigator — Centre for Medical Imaging
Locations (1):
- Centre for Medical Imaging, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes